CLINICAL TRIAL: NCT02619864
Title: A Phase I Study of the mTORC1/mTORC2 Kinase Inhibitor AZD2014 in Patients With Previously Treated Glioblastoma Multiforme
Brief Title: mTORC1/mTORC2 Kinase Inhibitor AZD2014 in Previously Treated Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I222
Record Dates: First submitted 2015-11-26; First posted 2015-12-02 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD2014 plus temozolomide (Experimental): Patients will receive single agent AZD2014 for 2 days immediately prior to surgery at a fixed dose of 125 mg bid po (i.e. on days -2, -1, and on morning of day 0 [day of surgery]). After recovery from surgery, patients will start the dose escalation (within 7-21 days after tumour resection).
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014

SUMMARY:
The standard or usual treatment for this disease is standard chemotherapy alone. AZD2014 is a new type of drug for glioblastoma multiforme. In the laboratory it has been shown to slow the growth of glioblastoma multiforme. In some animal studies AZD2014 seemed to work better when given with a drug called temozolomide.

DETAILED DESCRIPTION:
The purpose of this study is to find the highest dose of AZD2014 that can be tolerated without causing very severe side effects when receiving temozolomide and see what good and/or bad effects AZD2014 can have on the tumour. This is done by starting at a dose lower than the one that we know can be given safely to the participants when used on its own. Participants are given AZD2014 together with temozolomide and will be watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then new participants will be given a higher dose of AZD2014. Participants joining this study later on will get higher doses of AZD2014 than participants who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed glioblastoma multiforme that is recurrent after primary treatment (surgery/radiation/temozolomide) (i.e. first progression). Patients may not have had disease progression while receiving adjuvant temozolomide or radiation.
* All patients must have an available formalin fixed paraffin embedded tissue block (from their primary tumour) and must have provided informed consent for the release of the block. Patients participating in the pharmacodynamics study must have provided consent for release of a representative sample of the resected tumour.
* Presence of clinically and/or radiologically documented disease. MRI scan must be performed within 14 days prior to registration.
* All patients enrolled to DL3 and the dose expansion cohort at RP2D must have measurable disease according to RANO criteria as follows: At least one enhancing lesion which is ≥ 10 mm x 10 mm
* Patients must be ≥18 years of age.
* Patients must have an ECOG performance status of 0 or 1.
* Patients must have received one prior temozolomide regimen, discontinued at least 16 weeks prior to registration. Patients may have received one other cytotoxic regimen (for example CCNU).
* Patients may not have received immunotherapies, biologic and viral therapies, angiogenesis inhibitors, mTOR, or PARP inhibitors
* Patients must have recovered from all reversible toxicity related to prior chemotherapy and have adequate washout from prior chemotherapy, and investigational agents as follows: longest of one of the following:

  * two weeks,
  * standard cycle length of prior regimen,
  * 5 half-lives for investigational drugs.
* Prior external beam radiation must have been completed at least 4 weeks prior to registration.
* Previous surgery is permitted provided that a minimum of 21 days have elapsed between any major surgery (excluding resection for patients participating in the Pharmacodynamic Study) and date of registration, and that wound healing has occurred.
* Patients must have recovered from any treatment related toxicities prior to registration (unless grade 1, irreversible, or considered by investigator as not clinically significant).
* Hematology: Neutrophils ≥ 1.5 x 10^9/L; Platelets ≥ 100 x 10^9/L; INR ≤ 1.5
* Biochemistry:

Serum Creatinine or Creatinine Clearance* ≥ 50 ml/min (calculated by Cockcroft and Gault equation) Total bilirubin ≤ 1.5 x ULN AST and ALT ≤ 2.5 x ULN (≤ 5x ULN in the presence of liver metastases) Electrolytes within normal limits

* Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by appropriate formula below:

Females: GFR = 1.04 x (140-age) x weight in kg / serum creatinine in μmol/L

Males: GFR = 1.23 x (140-age) x weight in kg / serum creatinine in µmol/L

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate. Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.
* Patients must be accessible for treatment and follow up.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient registration (exceptions will be made if surgical resection is delayed).
* Women/men of childbearing potential must have agreed to use 2 methods of contraception (1 highly effective method and 1 barrrier method) until 4 weeks after the end of treatment. Acceptable methods of highly effective contraception include:

  * Placement of an intrauterine device or intrauterine system.
  * Male partner's sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
  * True abstinence.
  * Acceptable barrier methods of contraception include: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

Please note: use of oral, injected, or implanted hormonal methods of contraception cannot be considered highly effective as it is currently unknown whether AZD2014 may reduce their effectiveness).

Exclusion Criteria:

* Patients who have undergone any of the following procedures or experienced conditions currently or in the preceding 12 months:
* Coronary artery bypass graft
* Angioplasty
* Vascular stent
* Myocardial infarction (MI)
* Angina pectoris
* Congestive heart failure New York Heart Association (NYHA) Grade 2
* Ventricular arrhythmias requiring continuous therapy
* Supraventricular arrhythmias including atrial fibrillation, which are uncontrolled.
* Hemorrhagic or thrombotic stroke, including transient ischemic attacks or any other central nervous system bleeding
* Patients with a baseline LVEF ≤ 50% by MUGA scan, and ≤ 55% by ECHO.
* Patients with mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome or unexplained sudden death under 40 years of age.
* Any evidence of severe or uncontrolled systemic disease, active infection (including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or a prior history of tuberculosis), active bleeding or bleeding diathesis or renal diseases such as nephritis or renal tubular acidosis.
* Patients with history of pre-existing and/or clinically or radiologically active interstitial lung disease.
* History of hypersensitivity to protocol therapy or any excipient used in this study
* Patients who have significant gastrointestinal disease and who are unable to swallow capsules.
* Concurrent Medications
* Patients receiving other investigational agents.
* Patients receiving other anti-cancer agents, or radiation therapy.
* Patients receiving known QT/QTc-prolonging drugs.
* Co-medications which are moderate or potent inhibitors or inducers of CYP3A4/5 and CYP2C8, Pgp (MDR1) and BCRP or are sensitive or narrow therapeutic range substrates of the drug metabolizing enzymes CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters Pgp (MDR1), BCRP, OATP1B1, OATP1B3, OCT1 and OCT2 will be restricted. These should be discontinued prior to registration unless in the opinion of the investigator the risk/benefit is acceptable and no alternative medications are available (see Appendix V for washout periods).
* Patients taking corticosteroids must have been on a stable or decreasing dose for at least 14 days prior to registration.
* Patients who require oral anticoagulants should be switched to LMW heparin.
* Patients on enzyme inducing anticonvulsants.
* Patients who do not agree to avoid the ingestion of large amounts of grapefruit and Seville oranges (and other products containing these fruits, e.g. grapefruit juice or marmalade).
* Pregnant or lactating women. Women of childbearing potential must have a pregnancy test proven negative within 7 days prior to registration. Men and women of childbearing potential must agree to use adequate contraception
* Patients who do not agree to avoid excessive sun exposure and use adequate sunscreen protection while on study and for three months after.
* Patients with diabetes type I or uncontrolled type II as judged by the investigator.
* Patients with meningeal or extracranial GBM involvement.
* Live attenuated vaccination administered within 30 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of AZD2014 | Day 0

SECONDARY OUTCOMES:
Number and severity of adverse events | 30 months
Response rate per RANO criteria | 30 months
To evaluate the plasma levels of AZD2014 alone at the time of resection | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Warren Mason, Study Chair — Univ. Health Network-OCI/Princess Margaret Hospital, Toronto ON
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lapointe S, Mason W, MacNeil M, Harlos C, Tsang R, Sederias J, Luchman HA, Weiss S, Rossiter JP, Tu D, Seymour L, Smoragiewicz M. A phase I study of vistusertib (dual mTORC1/2 inhibitor) in patients with previously treated glioblastoma multiforme: a CCTG study. Invest New Drugs. 2020 Aug;38(4):1137-1144. doi: 10.1007/s10637-019-00875-4. Epub 2019 Nov 9. PMID 31707687